CLINICAL TRIAL: NCT03491332
Title: Effect of Heated Breathing Circuit on Intraoperative Core Temperature and Systemic Inflammation After Brain Surgery: a Prospective Randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1-2017-0087
Record Dates: First submitted 2018-03-08; First posted 2018-04-09 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Patients Scheduled for Brain Surgery
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group C (Placebo Comparator): general circuit group
  Interventions: Device: conventional circuit
- group H (Active Comparator): warm circuit group
  Interventions: Device: conventional humidification circuit
- group SH (Experimental): new warm circuit group
  Interventions: Device: new humidifaction heat circuit

INTERVENTIONS:
Device: conventional circuit — The patient enters the operating room without any pretreatment and attaches a standard patient monitoring device. Anesthesia was performed by intravenous anesthesia. After induction of anesthesia, alveolar recruitment is performed in supine position in all groups with 30 cmH2O for 5 seconds. Mechanical ventilator was set with tidal volume of 8 ml / kg, the inspiratory/ expiratory ratio of 1: 2 and respiratory rate was adjusted for targeting EtCO2 around 35mmHg. Keep the fresh air flow of the ventilator at 3 L / min and set the temperature to 37 ° C for the heating circuits of group H and group SH. An arterial cannulation and subclavian jugular vein catheter is inserted.
  The circuits were applied to each group as follows; conventional circuit or group C, conventional humidification circuit for group H and new humidification heat circuit for group SH, respectively. All other conditions were same among three groups.
  Other Names: group C for control group (n=39)
  Arms: group C
Device: conventional humidification circuit — The patient enters the operating room without any pretreatment and attaches a standard patient monitoring device. Anesthesia was performed by intravenous anesthesia. After induction of anesthesia, alveolar recruitment is performed in supine position in all groups with 30 cmH2O for 5 seconds. Mechanical ventilator was set with tidal volume of 8 ml / kg, the inspiratory/ expiratory ratio of 1: 2 and respiratory rate was adjusted for targeting EtCO2 around 35mmHg. Keep the fresh air flow of the ventilator at 3 L / min and set the temperature to 37 ° C for the heating circuits of group H and group SH. An arterial cannulation and subclavian jugular vein catheter is inserted.
  The circuits were applied to each group as follows; conventional circuit or group C, conventional humidification circuit for group H and new humidification heat circuit for group SH, respectively. All other conditions were same among three groups.
  Other Names: group H for conventional humidification circuit (n = 39)
  Arms: group H
Device: new humidifaction heat circuit — The patient enters the operating room without any pretreatment and attaches a standard patient monitoring device. Anesthesia was performed by intravenous anesthesia. After induction of anesthesia, alveolar recruitment is performed in supine position in all groups with 30 cmH2O for 5 seconds. Mechanical ventilator was set with tidal volume of 8 ml / kg, the inspiratory/ expiratory ratio of 1: 2 and respiratory rate was adjusted for targeting EtCO2 around 35mmHg. Keep the fresh air flow of the ventilator at 3 L / min and set the temperature to 37 ° C for the heating circuits of group H and group SH. An arterial cannulation and subclavian jugular vein catheter is inserted.
  The circuits were applied to each group as follows; conventional circuit or group C, conventional humidification circuit for group H and new humidification heat circuit for group SH, respectively. All other conditions were same among three groups.
  Other Names: group SH for new humidifaction heat circuit (n=39)
  Arms: group SH

SUMMARY:
Mechanical respiration during general anesthesia causes cold and dry gases to reach the lower airway, reduce the function of the airway mucosa, and cause accumulation of secretions. Inhaled dry gas is one of the causes of hypothermia during general anesthesia. To overcome this, the warm-humidifying breathing circuit uses warm, moisture-preserving gas to promote mucus mobility of the airway mucosal ciliate cells and prevents cold gases from evaporating from the mucosal surfaces which results lowering body temperature. We aimed to investigate the effect of newly developed Sohum warm humidifying respiration circuit (SH501) on the prevention of core body temperature reduction during surgery and systemic inflammation reaction.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 19
2. scheduled for brain surgery

Exclusion Criteria:

1. age < 19
2. patients with severe obstructive lung disease and/or restrictive lung disease patients
3. patients with infectious disease
4. surgery with prone position or lateral position
5. arrhythmia

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
core temperature | every 30 minute after induction of anesthesia until the end of anesthesia
upper airway temperature | every 30 minute after induction of anesthesia until the end of anesthesia
upper airway humidity | every 30 minute after induction of anesthesia until the end of anesthesia

SECONDARY OUTCOMES:
cytokine level | 1, 30, 60, 90, 120, 150, 180, 210, 240 minute after induction and 1 second after the operation
  pg/ml for Cytokine level(TNF-a, IL-1, IL-6, IL-8, IL-10)
dead space | every 30 minute after induction of anesthesia until the end of anesthesia
  % for Deadspace(Vd/Vt)
intrapulmonary shunt | every 30 minute after induction of anesthesia until the end of anesthesia
  Qs/Qt,
respiratory variables | every 30 minute after induction of anesthesia until the end of anesthesia
  mmHg for respiratory variables(PaO2, PaCO2, PvO2, PvCO2)
compliance | every 30 minute after induction of anesthesia until the end of anesthesia
  L/cmH2O for compliance(△V/△P)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No